CLINICAL TRIAL: NCT05740189
Title: Clinical Trial to Evaluate Safety and Efficacy of the C2 Cryoballoon 180° Ablation System for the Treatment of Dysplastic Barrett's Esophagus: CBAS180 De-escalation Study
Brief Title: CBAS180 De-escalation Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Koen Munters (Other)
Collaborators: Pentax Medical (Industry)
Responsible Party: Sponsor-Investigator, Koen Munters, Research Fellow, MD, Gastroenterology and Hepatology, St. Antonius Hospital
Organization: St. Antonius Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL73252.000.22
Record Dates: First submitted 2023-01-18; First posted 2023-02-22 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Barrett's Esophagus; Ablation Therapy; Cryotherapy; Cryoballoon Ablation
MeSH Terms: conditions — Barrett Esophagus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- C2 CryoBalloon 180 Ablation System (Experimental): C2 CryoBalloon 180 Ablation System will be used to ablate visible Barrett's esophagus
  Interventions: Device: C2 CryoBalloon 180° Ablation System

INTERVENTIONS:
Device: C2 CryoBalloon 180° Ablation System — The C2 CryoBalloon 180° Ablation System is a cryosurgical device with a nitrous oxide cooled balloon probe that is compatible with upper gastrointestinal therapeutic endoscopes.

SUMMARY:
Evaluate the efficacy and safety of the C2 CryoBalloon 180° Ablatie Systeem (CBAS180) at decremental doses for the treatment of dysplastic Barrett's epithelium.

DETAILED DESCRIPTION:
Cryoballoon ablation is a relatively new ablation technique for the treatment of dysplastic Barrett's esophagus (BE). Previous studies with this technique have shown that treatment is safe and effective. When compared to other ablation techniques, cryoballon ablation has several potential advantages, including less pain and less complications such as stricture formation after treatment. Recently, a cryoballoon ablation system has become available which enables treatment of larger esophageal surfaces. Although a recent clinical study with this new device has shown promising results, the lowest possible dose that optimally balances safety and efficacy is still unknown.

This study is a multicenter, prospective, intervention study consisting of two phases: the treatment phase and the follow-up phase.

During the treatment phase, patients will undergo an upper endoscopy during which CBAS180 treatment will be performed. Treatment consists of two CBAS180 applications, starting just below the gastroesophageal junction (GEJ), resulting in a circumferential ablation of 3cm in length. During the treatment phase, two doses will be tested consecutively starting with the lowest dose (i.e. 1.2mm/sec). For each dose a total of 25 patients will be included. An interim analysis will be performed after treatment of the first 25 patients with the lowest dose of 1.2mm/sec, before proceeding to treatment of the additional 25 patients with a higher dose of 1.1mm/sec.

The follow-up phase starts after CBAS180 treatment and ends after first follow-up endoscopy at 10 weeks (±2 weeks) after treatment. Therefore, the study duration will be approximately 3 months for each individual patient. The investigators expect to report the primary outcome for all participating patients within 2 years.

ELIGIBILITY:
Inclusion Criteria:

1. Flat type BE esophagus, with an indication for ablation therapy, defined as:

   1. Diagnosis of LGD or HGD in BE (confirmed by BE expert pathologist) or;
   2. Residual BE with any grade of dysplasia after endoscopic resection (by means of EMR or ESD) to treat non-flat BE, ≥6 weeks prior to enrolling the patient to this study. The ER pathology should indicate endoscopic treatment (i.e. only mucosal invasion or limited submucosal invasion (sm1), no lymphovascular infiltration, free vertical resection margins and not poorly differentiated).
2. Prague Classification Score of C≤3 and M≥1.
3. Patients should be ablation-naïve, meaning they have not undergone any previous endoscopic ablation therapy of the esophagus.
4. Older than 18 years of age at time of consent.
5. Fit for endoscopic therapy per institution's standards.
6. Provides written informed consent on the IRB-approved informed consent form.
7. Willing and able to comply with follow-up requirements.

Exclusion Criteria:

1. Esophageal stenosis preventing advancement of a therapeutic endoscope.
2. Any endoscopically visualized lesion such as ulcers, masses or nodules. Neoplastic nodules must first be treated with ER ≥6 weeks prior to planned treatment under this protocol.
3. Prior ER of >2cm in length and/or >50% of the esophageal lumen circumference.
4. History of locally advanced (>sm1) esophageal cancer.
5. History of esophageal varices.
6. Prior distal esophagectomy.
7. Active esophagitis LA grade B or higher.
8. Severe medical comorbidities precluding endoscopy.
9. Uncontrolled coagulopathy.
10. Pregnant or planning to become pregnant during period of study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2023-02-19 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2026-01-15 (Estimated)

PRIMARY OUTCOMES:
Efficacy: Dose response | 3 months
  Efficacy (dose response) will be evaluated by the BE surface regression percentage after 1 circumferential treatment session, as evaluated by the EGD-Adjudication Committee (EGD-AC) and confirmed by histological evidence of eradication of BE.
Safety: Incidence of Dose-related SAEs | 24hours
  Safety will be evaluated by the incidence of dose-related SAEs. Dose-related SAEs include pain in the treatment area greater than 6 (scored on a 0 to 10-point numeric rating scale (NRS)) at 24 hours post-treatment; symptomatic stricture requiring an additional EGD plus endoscopic dilation before first follow-up EGD; symptomatic stricture requiring endoscopic dilation at follow-up EGD; or any stricture (symptomatic or asymptomatic) preventing passage of the diagnostic endoscope at follow-up EGD.
Safety: Incidence of Dose-related SAEs | 7 days
  Safety will be evaluated by the incidence of dose-related SAEs. Dose-related SAEs include pain in the treatment area greater than 6 (scored on a 0 to 10-point numeric rating scale (NRS)) at 7 days post-treatment; symptomatic stricture requiring an additional EGD plus endoscopic dilation before first follow-up EGD; symptomatic stricture requiring endoscopic dilation at follow-up EGD; or any stricture (symptomatic or asymptomatic) preventing passage of the diagnostic endoscope at follow-up EGD.
Safety: Incidence of Dose-related SAEs | 30 days
  Safety will be evaluated by the incidence of dose-related SAEs. Dose-related SAEs include pain in the treatment area greater than 6 (scored on a 0 to 10-point numeric rating scale (NRS)) at 30 days post-treatment; symptomatic stricture requiring an additional EGD plus endoscopic dilation before first follow-up EGD; symptomatic stricture requiring endoscopic dilation at follow-up EGD; or any stricture (symptomatic or asymptomatic) preventing passage of the diagnostic endoscope at follow-up EGD.

SECONDARY OUTCOMES:
Feasibility: technical succes | Directly after procedure
  Feasibility (technical success) defined as the percentage of patients in whom all BE could be treated as intended by the treating endoscopist.
Post-procedural pain | Directly after procedure
  Post-procedure pain in the area of the cryoablation treatment (scored on a 0 to 10-point numeric rating scale (NRS)), described as the median pain score directly after treatment.
Post-procedural pain | 24 hours
  Post-procedure pain in the area of the cryoablation treatment (scored on a 0 to 10-point numeric rating scale (NRS)), described as the median pain score 1 day after treatment.
Post-procedural pain | 7 days
  Post-procedure pain in the area of the cryoablation treatment (scored on a 0 to 10-point numeric rating scale (NRS)), described as the median pain score 7 days after treatment.
Post-procedural pain | 30 days
  Post-procedure pain in the area of the cryoablation treatment (scored on a 0 to 10-point numeric rating scale (NRS)), described as the median pain score 30 days after treatment.
Post-procedure dysphagia | Directly after procedure
  Post-procedure dysphagia (scored on a 0-4 dysphagia score), described as the median dysphagia score directly after treatment.
Post-procedure dysphagia | 24 hours
  Post-procedure dysphagia (scored on a 0-4 dysphagia score), described as the median dysphagia score 1 day after treatment.
Post-procedure dysphagia | 7 days
  Post-procedure dysphagia (scored on a 0-4 dysphagia score), described as the median dysphagia score 7 days after treatment.
Post-procedure dysphagia | 30 days
  Post-procedure dysphagia (scored on a 0-4 dysphagia score), described as the median dysphagia score 30 days after treatment.
Incidence AE and SAE | 30 days
  Incidence of all serious and non-serious AEs up to 30 days post-treatment.
BE regression | 3 months
  BE surface regression percentage after 1 circumferential treatment session as assessed by the treating endoscopist.

CONTACTS AND LOCATIONS:
Locations (6):
- Netherlands (6):
  - Catharina Hospital, Eindhoven, North Brabant
  - Amsterdam UMC, Amsterdam, North Holland
  - UMC Groningen, Groningen, Provincie Groningen
  - Erasmus MC, Rotterdam, South Holland
  - St Antonius hospital, Nieuwegein, Utrecht
  - UMC Utrecht, Utrecht, Utrecht

IPD SHARING:
Plan to Share IPD: Undecided